CLINICAL TRIAL: NCT03125434
Title: Normative Dynamic & Magnetic Spine. Musculoskeletal Characteristics Static and Dynamic of Spine in Healthy Subject
Brief Title: Normative Dynamic & Magnetic Spine
Acronym: NDMS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: funding problems
Sponsor: Centre d'Investigation Clinique et Technologique 805 (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2016-A01825-46
Record Dates: First submitted 2017-03-21; First posted 2017-04-24 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Healthy Volunteers; Dynamic Stability Margin; Gait; Paraspinal Muscles
MeSH Terms: interventions — Magnetic Resonance Spectroscopy; Gait Analysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- healthy volunteers (Experimental): EOS full-spine, MRI, gait analysis
  Interventions: Other: EOS full-spine, MRI, gait analysis

INTERVENTIONS:
Other: EOS full-spine, MRI, gait analysis — full-spine stereoradiography, high-resolution spine muscle MRI and 3D gait analysis will be performed

SUMMARY:
This study aims to describe normal spinal musculoskeletal patterns in healthy adolescents and young adults by using static and dynamic measures. Static informations are obtained from full-spine stereoradiography for skeletal measures and from high-resolution spine muscle MRI for muscular data. Dynamics stability is calculated from 3D gait analysis.

DETAILED DESCRIPTION:
Spinal diseases and deformities in adults (degenerative or traumatic) and children (scoliosis and kyphosis) are major public health issues.

Postural imbalance due to spinal deformity is usually measured on static radiographs, using standard X-rays. However, bipedal walk is characteristic from human being and the trunk is the main stabilizer.

Pathogenesis of spinal deformities remains undefined. To understand the different mechanisms involved in the pathological field, normal musculoskeletal performances of the spine, in static and dynamic conditions must be identified.

Ultra-low doses stereoradiography using the EOS system allows the acquisition of full-spine images in standing position. Furthermore, 3D reconstruction can also be create from both anteroom-posterior and lateral side view. Stereoradiography is used in clinical routine especially in children spinal deformities.

High resolution muscular MRI is the only device that can provide a detailed muscular analysis, with detection of abnormalities at an early stage. No mapping of normal paraspinal muscles has been yet realized, particularly regarding to rotatores muscles.

Motion analysis is the reference exam to analyse dynamic stability during gait. Several parameters reflecting stability during gait can be collected in different conditions. Recently, the "Dynamic Stability Margin" has been developed but no standard values especially in healthy children has been published.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent signed by adult or by the holders of parental authority for the children and adolescents
* Child or teenager, male or female, aged from 8 years to 17 years inclusive
* Adult, male or female, aged from 18 years to 40 years inclusive
* Realization of a preliminary medical examination

Exclusion Criteria:

* Refuse to participate to the study
* Patient under guardianship or curatorship
* Inability to cooperate
* Pregnant woman
* Non affiliation to social security
* Subject with spinal and/or lower limbs affection
* Subject with antecedent of spinal and/or lower limbs surgery
* Subject with contraindication to MRI
* Refusal of the parent or the subject to be informed about a fortuitous discovery during the examinations of the exams

Ages: 8 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 48 (Actual)
Dates: Start 2017-04-27 (Actual); Primary Completion 2020-10-23 (Actual); Study Completion 2020-10-23 (Actual)

PRIMARY OUTCOMES:
Normal dynamic stability margin (DSM) in children and adults | 2 hours
  DSM= xCoM (extrapolated center of mass)- BoS (Base of Support). Unit = meters Normalized on body height (m)

SECONDARY OUTCOMES:
number of rotatores muscles | 2 hours
  counting every rotatore muscle (from MRI data), no unit
volume of back muscles | 2 hours
  from segmentation of each muscle group, unit = voxel

CONTACTS AND LOCATIONS:
Locations (1):
- APHP Hopital raymond Poincaré, Garches, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No